CLINICAL TRIAL: NCT02374177
Title: The Effects of Anaesthetic Agents on Postoperative Delirium in the Patients Undergoing Off-pump Coronary Artery Bypass Grafting Surgery
Brief Title: The Effects of Anaesthetic Agents on Postoperative Delirium
Status: Completed | Type: Observational
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: KUH1160073
Record Dates: First submitted 2015-02-04; First posted 2015-02-27 (Estimated); Last update posted 2015-02-27 (Estimated); Status verified 2015-02

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Propofol group: Patient anesthetized using propofol
- Sevoflurane group: Patients anesthetized using sevoflurane

SUMMARY:
The purpose of this study is to prove the correlation between the post-operative delirium (POD) and anesthetic agents. The investigators hypothesized that intravenous anaesthetics would show the lower incidence of POD, compared with inhalation anaesthetics in off-pump CABG.

DETAILED DESCRIPTION:
The medical records of the patients undergoing off-pump coronary artery bypass grafting (CABG) in Konkuk University Medical Centre from Jan 2010 to Aug 2014 were retrospectively reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing off-pump coronary artery bypass grafting

Exclusion Criteria:

* Other concurrent surgery
* Conversion from off-pump coronary artery bypass grafting to on-pump coronary artery bypass grafting

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The medical records of the patients undergoing off-pump CABG in Konkuk University Medical Centre from Jan 2010 to Aug 2014 were retrospectively reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | up to postoperative 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hyop Kim, Professor, Principal Investigator — Konkuk University Medical Center

REFERENCES:
- [Background] Koster S, Hensens AG, van der Palen J. The long-term cognitive and functional outcomes of postoperative delirium after cardiac surgery. Ann Thorac Surg. 2009 May;87(5):1469-74. doi: 10.1016/j.athoracsur.2009.02.080. PMID 19379886